CLINICAL TRIAL: NCT01286584
Title: Smoking Cessation in a Drug Treatment Program: A Randomized Trial of Varenicline Versus Placebo.
Brief Title: Varenicline in Drug Treatment
Acronym: ViRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 144/2010-02
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Smoking Cessation; Alcohol Abuse
Keywords: varenicline; alcohol; placebo; smoking cessation
MeSH Terms: conditions — Smoking Cessation; Alcoholism | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- varenicline group (Active Comparator)
  Interventions: Drug: varenicline
- placebo group (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — one 0.5mg varenicline capsule on first 3 days one 0.5mg varenicline capsule, twice daily for 4 days one 1.0mg varenicline capsule, twice daily until end of treatment (12weeks of medication
  Other Names: Champix; Chantix
  Arms: varenicline group
Drug: placebo — lactose filler in capsules identical to the varenicline capsules one 0.5mg capsule for 3 days one 0.5mg capsule twice daily for 4 days one 1.0mg capsule twice daily until end of treatment (12weeks of medication)
  Arms: placebo group

SUMMARY:
The aim of this study is to assess the efficacy of varenicline compared to placebo in tobacco dependent individuals who are undergoing concurrent treatment for alcohol dependence. As they will be inpatients and under 24 hour medical care for the first 21 days of treatment, or receiving outpatient treatment through the Alcohol Research and Treatment Clinic, this will allow for a comprehensive assessment of the safety of varenicline in this population with minimal risk of adverse consequences. The patients will continue their cessation treatment for an additional 10 weeks as outpatients through the Nicotine Dependence Clinic at CAMH. They will also be contacted at 6 months for follow-up.

DETAILED DESCRIPTION:
Drinking alcohol and cigarette smoking are closely associated and use of one often leads to the use of the other. Also, since tobacco-related illness is the number one cause of death among recovered alcoholics it is imperative that we provide strong evidence-based treatment options for this population. Since smoking can be a strong trigger to drink in those who are dependent on both alcohol and tobacco, treating both at the same time may result in better treatment outcomes. This study will examine the efficacy of starting smoking cessation treatment while patients are in residential treatment for alcohol dependence, or outpatient in the Alcohol Research and Treatment Clinic. It will compare the effectiveness of varenicline, the most effective medication for smoking cessation with placebo. Both groups will receive weekly cessation counselling and support by a trained research analyst. We will measure abstinence from smoking at the end of the 12-week treatment period and again after 6-months to determine longer-term smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* current daily smokers enrolled in residential treatment or outpatient in Alcohol Treatment and Research Clinic for Alcohol Use Disorder at CAMH
* smoke minimum of 10 cigarettes per day
* Fagerstrom Test of Nicotine Dependence score > 3
* able to provide written informed consent
* able and willing to attend weekly appointments at the NDC following discharge

Exclusion Criteria:

* any serious medical condition requiring immediate investigation or treatment
* pregnancy or lactation
* current DSM-IV Axis I psychiatric disorder
* any know contraindication to using varenicline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
quit smoking rating | end of 12-week treatment
  7-day point prevalence

SECONDARY OUTCOMES:
30 day continuous smoking abstinence | 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Nicotine Dependence Clinic, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research